CLINICAL TRIAL: NCT01943084
Title: A Trial to Investigate the Bioequivalence of Norditropin® (Somatropin) Versus Genotropin® (Somatropin) in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GH-4108; U1111-1143-0754 (Other: WHO)
Record Dates: First submitted 2013-09-10; First posted 2013-09-16 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-01

CONDITIONS: Growth Disorder; Healthy
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Norditropin® (Experimental)
  Interventions: Drug: Norditropin® FlexPro® pen
- Genotropin® (Active Comparator)
  Interventions: Drug: Genotropin Pen®

INTERVENTIONS:
Drug: Norditropin® FlexPro® pen — Administered as a single subcutaneous (s.c., under the skin) dose (4.0 mg) on 2 separate dosing visits (treatment periods). The 2 treatment periods will be separated by a 7-day washout period.
  Arms: Norditropin®
Drug: Genotropin Pen® — Administered as a single subcutaneous dose (4.0 mg) on 2 separate dosing visits (treatment periods). The 2 treatment periods will be separated by a 7-day washout period.
  Arms: Genotropin®

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of the trial is to investigate the bioequivalence (the expected biological equivalence of two pharmaceutical drug products with identical active ingredient) of Norditropin® (somatropin) versus Genotropin® (somatropin) in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects at trial entry with no previous exposure to recombinant human growth hormone or IGF-I (insulin-like growth factor-I)
* Body mass index (BMI) 18.0-27.0 kg/m^2 (both inclusive)
* Considered generally healthy upon completion of medical history, physical examination, vital signs, screening laboratory results, and electrocardiogram (ECG), as judged by the investigator

Exclusion Criteria:

* The receipt of any investigational medicinal product within 1 month prior to this trial
* Current or previous treatment with growth hormone or IGF-I
* Female of childbearing potential who is pregnant, breast-feeding or intends to become pregnant or is not using adequate contraceptive methods (adequate contraceptive measures as required by local law or practice) for the duration of the trial
* Known presence or history of malignancy
* Diabetes mellitus
* Use of systemic corticosteroids
* Use of anabolic steroids
* History of drug or alcohol abuse

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Area under the serum hGH (human growth hormone) concentration-time curve | From 0 to the time of the last quantifiable concentration over a 24-hour sampling period.
Maximum observed serum hGH concentration | Over a 24-hour sampling period
Area under the effect (IGF-I) (insulin-like growth factor-I) curve | From time 0 to the time of the last measurable concentration (AUEC0-t) (area under the effect curve) over a 96-hour sampling period
Maximum IGF-I effect (Emax) | Over a 96-hour sampling period

SECONDARY OUTCOMES:
The frequency of adverse events (AE) | From screening to follow-up period (up to day 23)
Abnormal haematology laboratory parameters | From screening to follow-up period (up to day 23)
Abnormal biochemistry laboratory parameters | From screening to follow-up period (up to day 23)
The frequency of injection-site reactions | From the time of injection of the trial product to follow-up during the 2 dosing periods (on Days 1 through 5, with visit 7 as follow-up and separately on Days 13 through 17, with visit 12 as follow-up for each period)
Area under the effect (IGFBP-3) (insulin-like growth factor binding protein 3) curve | From time 0 to the time of the last concentration (AUEC0-t) over a 96-hour sampling period
Maximum IGFBP-3 effect (Emax) | Over a 96-hour sampling period
Abnormal findings in vital signs | From screening to follow-up period (up to day 23)
Abnormal findings in physical examinations | From screening to follow-up period (up to day

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Clinical Trial Call Center, Overland Park, Kansas, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com